CLINICAL TRIAL: NCT04032743
Title: Retrospective Study: Risk Factors and Treatment Outcome of Oncology Children Hospitalized in the Intensive Care Unit Due to Sepsis
Brief Title: Risk Factors and Treatment Outcome of Oncology Children Hospitalized in the Intensive Care Unit Due to Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0590-18-RMC
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Oncologic Complications and Emergencies; ICU; Sepsis; Childhood Cancer
MeSH Terms: conditions — Emergencies; Sepsis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ICU treatment — any treatment available by ICU

SUMMARY:
Children treated with intensive chemotherapy are at increased risk for life-threatening infections (sepsis). As the survival of oncology patients increased with the use of aggressive treatment protocols, there was also an increase in the need for hospitalization in intensive care units (ICU) due to sepsis.Several prognostic factors are known to affect the survival of these patients, including the number and type of damaged systems, the type of oncology disease and the duration of neutropenia. With the development of the treatment of ICU, the survival of the oncology patients hospitalized for sepsis has also increased.

We will collect demographic details, details of their oncology and infections, laboratory tests and imaging. The goal is to identify prognostic factors in oncologic children hospitalized in ICU due to sepsis, as well as clinical and laboratory parameters that characterize this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Treatment in the hemato-oncology for cancer
* Admission to the ICU in SCMCI between 2008-2018 because of sepsis during chemotherapy

Exclusion Criteria:

* Admission to the ICU more than 3 month after last chemotherapy or 1 year after SCT

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and youth treated at Schneider Children's Hospital with chemotherapy due to oncology and hospitalized at Schneider Children's Hospital from 2008 until the end of 2018 due to sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
survival | 30 day
  survial status 30 day after release from the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Barzilai Birenboim, MD, Principal Investigator — Schneider Children's Medical Center in Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Specific requests for collaborative work and IPD sharing will be considered upon request.